CLINICAL TRIAL: NCT00655473
Title: A Randomized, Placebo-controlled Study of the Effect of RO4607381 on Progression or Regression of Atherosclerotic Plaque in Patients With Coronary Heart Disease (CHD) Including Patients With Other CHD Risk Factors
Brief Title: A Study of the Effect of RO4607381 on Atherosclerotic Plaque in Patients With Coronary Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NC21153
Record Dates: First submitted 2008-03-28; First posted 2008-04-10 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — dalcetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dalcetrapib (RO4607381) (Experimental)
  Interventions: Drug: Dalcetrapib (RO4607381)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dalcetrapib (RO4607381) — 600mg po daily for 24 months
  Arms: Dalcetrapib (RO4607381)
Drug: Placebo — po daily for 24 months
  Arms: Placebo

SUMMARY:
This study will assess the effect of RO4607381, compared to placebo, on atherosclerotic plaque in patients with coronary heart disease (CHD) including patients with other CHD risk factors. After a pre-randomisation period during which positron emission tomography computed tomography (PET/CT) and MRI will be conducted, patients will be randomized to receive either RO4607381 600mg po daily, or placebo po daily. PET/CT and MRI scans will be taken at intervals during the study. The anticipated time on study treatment is 2 years, and the target sample size is 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* CHD, including patients with other CHD risk factors;
* treated appropriately for dyslipidemia;
* clinically stable.

Exclusion Criteria:

* previous exposure to any cholesteryl ester transfer protein (CETP) inhibitor or vaccine;
* recent (within 3 months) clinically significant coronary events, transient ischemic attacks or cerebrovascular accident;
* severe anemia;
* uncontrolled hypertension;
* poorly controlled diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- United States (10):
  - Jacksonville, Florida
  - Royal Oak, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - New York, New York
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Houston, Texas
  - Seattle, Washington
- Montreal, Quebec, Canada

REFERENCES:
- [Derived] Duivenvoorden R, Mani V, Woodward M, Kallend D, Suchankova G, Fuster V, Rudd JHF, Tawakol A, Farkouh ME, Fayad ZA. Relationship of serum inflammatory biomarkers with plaque inflammation assessed by FDG PET/CT: the dal-PLAQUE study. JACC Cardiovasc Imaging. 2013 Oct;6(10):1087-1094. doi: 10.1016/j.jcmg.2013.03.009. PMID 24135322
- [Derived] Calcagno C, Ramachandran S, Izquierdo-Garcia D, Mani V, Millon A, Rosenbaum D, Tawakol A, Woodward M, Bucerius J, Moshier E, Godbold J, Kallend D, Farkouh ME, Fuster V, Rudd JH, Fayad ZA. The complementary roles of dynamic contrast-enhanced MRI and 18F-fluorodeoxyglucose PET/CT for imaging of carotid atherosclerosis. Eur J Nucl Med Mol Imaging. 2013 Dec;40(12):1884-93. doi: 10.1007/s00259-013-2518-4. Epub 2013 Aug 14. PMID 23942908
- [Derived] Fayad ZA, Mani V, Woodward M, Kallend D, Abt M, Burgess T, Fuster V, Ballantyne CM, Stein EA, Tardif JC, Rudd JH, Farkouh ME, Tawakol A; dal-PLAQUE Investigators. Safety and efficacy of dalcetrapib on atherosclerotic disease using novel non-invasive multimodality imaging (dal-PLAQUE): a randomised clinical trial. Lancet. 2011 Oct 29;378(9802):1547-59. doi: 10.1016/S0140-6736(11)61383-4. Epub 2011 Sep 9. PMID 21908036

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Started | 64 | 66
Completed | 53 | 51
Not Completed | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalcetrapib (RO4607381) | Placebo | Total
Number analyzed (Participants) | 64 | 66 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.24) | 64.6 (7.8) | 63.6 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 55 | 106
  Male | 13 | 11 | 24
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 8 | 16
  United States | 56 | 58 | 114

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Mean Wall Thickness
Time Frame: 24 months
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 64 | 66
Percent Change | 4.245 (3.018) | 6.679 (3.111)

2. Primary Outcome: Change From Baseline in Target (Plaque) to Background (Blood) Ratio From an Index Vessel.
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 64 | 66
Ratio | -0.188 (0.078) | -0.260 (0.079)

3. Secondary Outcome: Change From Baseline in Vessel Magnetic Resonance (MR) Determined Compliance
Time Frame: 6 months
Population: Data not collected
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Vessel MR Determined Plaque Anatomy
Time Frame: Up to 24 months
Population: Data not collected
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Blood Lipids,Lipoproteins
Time Frame: Throughout study
Population: Data not collected
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Biomarkers
Time Frame: Up to 24 months
Population: Data not collected
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: CHD, Major Coronary Events, Adverse Events (AEs), Lab Parameters, Blood Pressure
Time Frame: Throughout study
Population: Data not collected
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Serious Adverse Events (participants affected / at risk) | 20/64 | 19/66
Other Adverse Events (participants affected / at risk) | 0/64 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalcetrapib (RO4607381) (N=64) | Placebo (N=66)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Scrotal Abcess (Infections and infestations) | 1 (1) | 0 (0)
Scrotal Infection (Infections and infestations) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 3 (3)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Stent-Graft Endoleak (General disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No